CLINICAL TRIAL: NCT06064123
Title: Biomarkers for Diagnosis, Prognosis, and Targeted Therapy After Heart Transplantation
Acronym: EMBIO
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Helsinki University Central Hospital (Other)
Responsible Party: Principal Investigator, Karl Lemstrom, Professor of Cardiothoracic surgery, Helsinki University Central Hospital
Other Study IDs: HUS/3654/2017
Record Dates: First submitted 2023-06-20; First posted 2023-10-03 (Actual); Last update posted 2023-10-03 (Actual); Status verified 2023-10

CONDITIONS: Heart Transplant Rejection
Keywords: Donor-derived Cell-Free DNA; Platelet; Endomyocardial biopsy; Liquid biopsy; Transcriptome; Proteomics; Metabolomics; Glycoproteins; Surveillance; Extracellular Vesicles
MeSH Terms: interventions — Noninvasive Prenatal Testing

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples With DNA — Endomyocardial biopsies, peripheral blood platelets, peripheral blood extracellular vesicles, peripheral blood leukocytes, peripheral blood plasma, peripheral blood cell-free DNA, proteomics, metabolomics, glycoproteins
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cardiac transplant recipients: The group consist of all recruited cardiac transplant recipients operated in Helsinki University Hospital
  Interventions: Diagnostic Test: Cell-free DNA

INTERVENTIONS:
Diagnostic Test: Cell-free DNA — Donor-derived cell-free DNA relation to recipient-derived cell-free DNA is compared to histopathological rejection grade from the same time frame.

SUMMARY:
The objective of this prospective observational single center study is to investigate donor-derived cell-free DNA (ddcfDNA), peripheral blood platelet mRNA, peripheral blood extracellular vesicle mRNA, and peripheral blood leukocyte mRNA expression in recognition of clinically significant endomyocardial biopsy (EMB) proven acute rejection in human heart transplant recipients. In detail, the objective is to develop novel biomarkers and liquid biopsies for diagnosis, prognosis, and targeted molecular therapy for primary graft failure, ischemia-reperfusion injury, acute rejection, and development of late graft failure and cardiac allograft vasculopathy, and for monitoring immunosuppression after heart transplantation.

ELIGIBILITY:
Inclusion Criteria:

* patient age > 18 years
* heart transplant recipient
* has signed informed consent

Exclusion Criteria:

* foreign residency
* no signed informed consent collected

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Study population consist of heart transplant recipients transplanted at the Helsinki University Hospital, Helsinki, Finland.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2019-01-22 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Plasma donor-derived cell-free DNA (dd-cfDNA) for routine surveillance of acute rejection after heart transplantation | 5 years
  To compare plasma dd-cfDNA to endomyocardial biopsy data
Allograft educated platelet-derived mRNA for gene expression profiling of acute rejection after heart transplantation | 5 years
  To compare gene expression profile of allograft-educated platelets to endomyocardial biopsy data
Plasma extracellular vesicle (EV) derived mRNA for gene expression profiling of acute rejection after heart transplantation | 5 years
  To compare gene expression profile of EV-derived mRNA to endomyocardial biopsy data
Plasma glycoproteins for routine surveillance of acute rejection after heart transplantation | 5 years
  To compare plasma glycoproteome profile to endomyocardial biopsy data

SECONDARY OUTCOMES:
Plasma metabolomics changes during acute rejection after heart transplantation | 1 year
  Plasma metabolic changes will be measured by mass spectrometry during routine surveillance endomyocardial biopsies taken at 2, 4, 6, 8, and 12 weeks and at 4, 5, 6, 8, 10, and 12 months after heart transplantation to investigate if there are any plasma metabolomics changes during different grades of acute rejection.
Plasma proteomics changes during acute rejection after heart transplantation | 1 year
  Plasma proteomics changes will be measured by mass spectrometry during routine surveillance endomyocardial biopsies taken at 2, 4, 6, 8, and 12 weeks and at 4, 5, 6, 8, 10, and 12 months after heart transplantation to investigate if there are any plasma proteomics changes during different grades of acute rejection during the first year.
Peripheral blood mononuclear cell mRNA expression for gene expression profiling of acute rejection after heart transplantation | 1 year
  To compare gene expression profile of peripheral blood mononuclear cells to endomyocardial biopsy data
Plasma metabolomics changes during the first year after heart transplantation and their relationship to the development of cardiac allograft vasculopathy | 5 years
  Plasma metabolomics changes will be measured by mass spectrometry during routine surveillance endomyocardial biopsies taken at 2, 4, 6, 8, and 12 weeks and at 4, 5, 6, 8, 10, and 12 months after heart transplantation and their relationship to the development of cardiac allograft vasculopathy in coronary angiogram will be investigated at 1, 3, and 5 years.
Plasma metabolomics changes during the first year after heart transplantation and their relationship to patient survival at 1, 3, and 5 years | 5 years
  Plasma metabolomics changes will be measured by mass spectrometry during routine surveillance endomyocardial biopsies taken at 2, 4, 6, 8, and 12 weeks and at 4, 5, 6, 8, 10, and 12 months after heart transplantation and their relationship to patient survival will be investigated at 1, 3, and 5 years.
Plasma proteomics changes during the first year after heart transplantation and their relationship to the development of cardiac allograft vasculopathy | 5 years
  Plasma proteomics changes will be measured by mass spectrometry during routine surveillance endomyocardial biopsies taken at 2, 4, 6, 8, and 12 weeks and at 4, 5, 6, 8, 10, and 12 months after heart transplantation and their relationship to the development of cardiac allograft vasculopathy in coronary angiogram will be investigated at 1, 3, and 5 years.
Plasma proteomics changes during the first year after heart transplantation and their relationship to patient survival at 1, 3, and 5 years | 5 years
  Plasma proteomics changes will be measured by mass spectrometry during routine surveillance endomyocardial biopsies taken at 2, 4, 6, 8, and 12 weeks and at 4, 5, 6, 8, 10, and 12 months after heart transplantation and and their relationship to patient survival will be investigated at 1, 3, and 5 years.

CONTACTS AND LOCATIONS:
Overall Officials: Karl B Lemström, MD, PhD, Principal Investigator — Helsinki University Central Hospital
Locations (1):
- Helsinki University Hospital, Helsinki, Uusimaa, Finland

IPD SHARING:
Plan to Share IPD: Undecided